CLINICAL TRIAL: NCT01938859
Title: Algorithm Guided Treatment Strategies for Bipolar Depression
Acronym: AGTs-BD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Yiru FANG M.D., Ph.D., M.D., Ph.D., Professor of Psychiatry, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012BAI01B04-BD; 2012BAI01B04 (Other Grant/Funding Number: 2012BAI01B04)
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; lithium; quetiapine; Medicine, Chinese Traditional; efficacy; safety; Recurrence
MeSH Terms: conditions — Bipolar Disorder; Recurrence | interventions — Lithium; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lithium combined with SGAs (Experimental): SGAs (Second Generation Antipsychotics), quetiapine adjunctive to lithium therapy
  Interventions: Drug: Lithium; Drug: Quetiapine
- lithium combined with TCM (Experimental): TCM (Traditional Chinese Medicine), Shuganjieyu capsule adjunctive to lithium therapy.
  Interventions: Drug: Lithium; Drug: Shuganjieyu capsule
- Lithium monotherpy (Active Comparator): Lithium monotherapy
  Interventions: Drug: Lithium

INTERVENTIONS:
Drug: Lithium — Lithium plasma concentration was between 0.6-1.2 mmol/L, dose should be fixed at the end of week 4, and the maximum dosage was judged by the investigator based on the patients' tolerability.
Drug: Quetiapine — Quetiapine adjunctively to lithium therapy, target 400 mg/d with a minimum dose of 200 mg/d. Dose should be fixed at the end of week 4, and the maximum dosage was judged by the investigator based on the patients' tolerability.
  Arms: Lithium combined with SGAs
Drug: Shuganjieyu capsule — Shuganjieyu capsule adjunctively to lithium therapy, target dose 1440 mg/d.
  Other Names: SGJY, St.John's wort and acanthopanax senticosus combination
  Arms: lithium combined with TCM

SUMMARY:
The purpose of the AGTs-BD study is to compare the treatment outcome and safety profiles between different mood stabilizers combination treatments in the patients with bipolar disorders, currently suffered from depression episode.

DETAILED DESCRIPTION:
The AGTs-BD study is a randomized, open-label, rater-blind, multicenter study, which including an 8-week acute treatment (Phase I), followed by a 24-week recurrence prevention treatment (Phase II), and a 24-week relapse prevention treatment (Phase III). Patients initially enter an up to 4 weeks screening phase to confirm the randomization to whom met DSM-IV criteria of bipolar I or II disorder, currently depressed with Hamilton Depression Rating Scale-17 items (HAM-D) total score ≥17. The protocol was approved by the each sites' appropriate institutional review boards and ethics committees. After screening, patients were randomly allocated to one of three groups: (1) lithium monotherapy; (2) lithium plus quetiapine; (3) lithium plus a Traditional Chinese Medicine (TCM) named as Shuganjieyu capsule (SGJY, St. John's wort and acanthopanax senticosus combination). After phase I, patients who met stable remission, defined as HAM-D total score ≤7 and Young Mania Rating Scale (YMRS) total score ≤10 in two consecutive visit at least 4 weeks, were qualified into phase II and III. Patients remained on the allocated treatment for up to 48 weeks or until treatment failure. The difference between phase II and phase III was that treatment dose could be decreased (within the study ranges) if side-effects became troublesome in phase III, but not for phase II. All patients will be provided with free care (3 visits) by the investigators, for a period of up to 3 months after the end of the study, in order to help them make the transition into routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old;
* Han Chinese;
* Outpatient and inpatient patients;
* Patients met DSM-IV criteria of bipolar I or II disorder, currently depressed, ascertained with the Mini International Neuropsychiatric Interview (MINI)
* HAM-D total score≥17, HAM-D item 1 (depressed mood) score≥2, and YMRS total score≤10 at baseline;
* Written informed consent was given;
* Junior high school education and above, with enough audio-visual ability to accomplish the visits;
* Normally resident in one country and had a residential address, able to follow-up.

Exclusion Criteria:

* Bipolar disorder rapid cycling or mixed episode;
* Experienced DSM-IV-TR axis I disorders in the 6 months prior to randomization;
* Severe personality disorder, metal retardation, anorexia/bulimia nervosa;
* Actively suicide ascertained by research psychiatrist or HAM-D item 3 score≥3(suicidality);
* Known history of intolerance or hypersensitivity to any of the medications involved in the study, including lithium, quetiapine and SGJY capsule;
* Female patients who were pregnant, planning to be pregnant or breast feeding;
* Severe medical or neurological problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The change of HAM-D total score only for the phase I | baseline and 8 weeks
Time to new intervention for an emerging mood episode | up to 48 weeks
  Time to new intervention for an emerging mood episode is only for Phase II and Phase III, including drug treatment (commencement of a new drug, increase in dose of concurrent drug, restarting of a discontinued drug, or increasing the investigational drug dose in response to an emergent mood episode) or admission to hospital.

SECONDARY OUTCOMES:
HAM-D total score ≤7 | 8 weeks for phase I, up to 48 weeks for phase II and III
  Remission rate
Mean changes from baseline to EOS in HAM-D total score ≥50% | 8 weeks for phase I, up to 48 weeks for phase II and III
  Response rate
Mean changes from baseline to EOS in 16-item Quick Inventory of Depressive Symptomatology-Patient Self-Report (QIDS16-SR) | 8 weeks for phase I, up to 48 weeks for phase II and III
Mean changes from baseline to EOS in Clinical Global Impression scale of Bipolar Disorder-Severity (CGI-BP-S) | 8 weeks for phase I, up to 48 weeks for phase II and III
Mean changes from baseline to EOS in Sheehan Disability Scale (SDS) | 8 weeks for phase I, up to 48 weeks for phase II and III
  Social function
Mean changes from baseline to EOS in 6-item Quality of Life scale (QOL-6) | 8 weeks for phase I, up to 48 weeks for phase II and III
  Social function
Young Mania Rating Scale (YMRS) total score ≤10 | 8 weeks for phase I, up to 48 weeks for phase II and III
  Using YMRS total score to monitor the switching from depression to hypomania and mania

CONTACTS AND LOCATIONS:
Overall Officials: Yiru Fang, M.D., Ph.D., Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China